CLINICAL TRIAL: NCT05021809
Title: Assessment of Postoperative Pain After Using Two Formulations of Calcium Hydroxide Intracanal Medication : A Randomized Clinical Trial.
Brief Title: Assessment of Postoperative Pain After Using Two Formulations of Calcium Hydroxide Intracanal Medication .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Sarah Alaa El Din Mohamed Hamed El Abyad, demonstrator at endodontic department, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 360/2021
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Necrotic Pulp With Symptomatic Apical Periodontitis
Keywords: pulp necrosis; symptomatic apical periodontitis; calcium hydroxide intracanal medication; postoperative pain; calcium hydroxide with iodoform; calcium hydroxide without iodoform
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blind allocation will be followed in the study .
  * Group A: will not receive any intracanal medication.(control group)
  * Group B :will recieve calcium hydroxide intracanal medication without iodoform (Metapaste)
  * Group c: will receive calcium hydroxide intracanal medication with iodoform (Metapex).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (No Intervention): control group will not receive any intracanal medication
- Group B (Active Comparator): Calcium hydroxide intracanal medication without iodoform (Metapaste )
  Interventions: Drug: Calcium hydroxide intracanal medication application
- Group C (Active Comparator): Calcium hydroxide intracanal medication with iodoform (Metapex)
  Interventions: Drug: Calcium hydroxide intracanal medication application

INTERVENTIONS:
Drug: Calcium hydroxide intracanal medication application — The patient will be anaesthized with Articaine hydrochloride 40 mg/ml + 1/100000 Epinephrine bitartrate solution . Then the rubber dam isolation will be conducted, the access will be opened and then cleaning and shaping will be done by using Protaper Next rotary file system and irrigation by sodium hypochlorite 2.5% by side vented needle, EDTA 17%, sodium hypochlorite and the final rinse by saline where the canal will be dried by absorbent paper point. The application of calcium hydroxide intracanal medication will be done according to the manufacturer instructions then temporization by glass ionomer will be applied .
  Arms: Group B; Group C

SUMMARY:
Calcium hydroxide is advocated as an intracanal medication for various purposes, including prevention of post-treatment symptoms. Calcium hydroxide has a pain-controlling effect at different times when compared to non-intracanal medication .

Aim:

The aim of the study to compare between postoperative pain after using two formulations of calcium hydroxide intracanal medication with and without iodoform .

DETAILED DESCRIPTION:
The most persuasive factor for a patient to visit a dental health care professional is the existence of odontalgia. Accordingly, the pain after a dental therapy results in demotivation of the patient. Unfortunately, mild to severe pain following a tooth-preserving therapy such as root canal treatment is reported to be experienced by 40% of the patients.

The majority of patients with symptomatic necrotic teeth had significant postoperative pain and required analgesic medication to manage this pain.

There is a correlation between the intensity of preoperative pain and postoperative pain ,The preoperative pain has a significant influence on postoperative pain.

Several strategies are suggested to manage or prevent post instrumentation pain. One of them is insertion of intracanal medicament.

The interappointment intracanal medicaments are suggested for disinfection of the infected root canal system in multi-visit endodontic treatment. Calcium hydroxide (Ca(OH)2) is considered as a universal intracanal medicament for this purpose.

Additionally, calcium hydroxide is hypothesized to exert a pain-preventing effect indirectly through its antimicrobial and tissue modifying properties .

Significantly high healing rates have been shown with short term use of calcium hydroxide Ca(OH)2 in teeth with apical periodontitis. As a temporary root filling, it has been shown to be an effective antimicrobial agent when applied for a minimum of 1 week.

Calcium hydroxide is a suitable material of choice as an inter-appointment dressing for teeth diagnosed with pulpal necrosis and apical periodontitis.

Calcium hydroxide reduced pain risk than no intracanal medication within the 1-14 days interval as well as triple-antibiotic paste within the first day and was similar to corticosteroid/antibiotics combination.

Iodoform has bacteriostatic property by releasing free iodine.Thereby, iodine eliminates the infection of root canal and periapical tissue by precipitating protein and oxidizes essential enzymes.

The use of calcium hydroxide-iodoform-silicon-oil paste as nonsurgical approach for treatment of periapical lesions showed a high success rate.

As clinicians , one of the most important goals to achieve is reducing the pain of the patient. Up to our knowledge, none of the previous studies investigated the postoperative pain incidence after application of Ca(OH)2 with iodoform as an intracanal medication .

ELIGIBILITY:
Inclusion Criteria:

* .single-rooted teeth with pulpal necrosis and symptomatic apical periodontitis with visible radiographic disturbance of periapical lamina dura. The diagnosis of pulp necrosis was confirmed by negative response to cold test, electric pulp tester and clinically by absence of blood upon access cavity .
* Clinical signs of apical periodontitis.
* Teeth with sufficient coronal tooth structure for adequate rubber dam isolation were selected .
* Patients who are over 18 years old .

Exclusion Criteria:

* Presence of open apices
* Presence of non-restorable teeth
* Presence of large carious lesions approaching the root.
* Presence of calcification or resorption .
* Patients who had received antibiotics during the last 3 months .
* Teeth with periodontal probing depth > 4 ml.
* Teeth with previous root canal treatment .
* Teeth with fluctuant facial swelling .
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 4 hours .
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 4 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 6 hours.
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 6 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 12 hours .
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 12 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 24 hours .
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 24 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 48 hours .
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 48 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded at 72 hours .
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded at 72 hours . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.
Measuring the severity of postoperative pain in both groups. | The pain score will be recorded after one week.
  Measuring the severity of postoperative pain in both groups. The patients will be informed to record their pain scores in visual analogue scale (VAS) as used by Habib et al. (1990) .The degree of the pain will have numerical value 0= no pain, 1-3= mild pain, 4-6= moderate pain , 7-9= severe pain . The pain score will be recorded after one week . No medication will be prescribed for the patients . They will be instructed to take only Ibuprofen if they experienced pain and it will be recorded in the chart.

CONTACTS AND LOCATIONS:
Overall Officials: marwa es sharaan, PHD, Principal Investigator — Suez Canal University
Locations (1):
- Endodontic Clinic At Faculty of Dentistry ,Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet

REFERENCES:
- [Background] Walton RE, Holton IF Jr, Michelich R. Calcium hydroxide as an intracanal medication: effect on posttreatment pain. J Endod. 2003 Oct;29(10):627-9. doi: 10.1097/00004770-200310000-00003. PMID 14606782
- [Background] Sebastian R, Drum M, Reader A, Nusstein J, Fowler S, Beck M. What is the Effect of No Endodontic Debridement on Postoperative Pain for Symptomatic Teeth with Pulpal Necrosis? J Endod. 2016 Mar;42(3):378-82. doi: 10.1016/j.joen.2015.12.001. Epub 2016 Jan 20. PMID 26806591
- [Background] Madarati AA, Zafar MS, Sammani AMN, Mandorah AO, Bani-Younes HA. Preference and usage of intracanal medications during endodontic treatment. Saudi Med J. 2017 Jul;38(7):755-763. doi: 10.15537/smj.2017.7.18345. PMID 28674723